CLINICAL TRIAL: NCT04812574
Title: Periurethral Hypertonic Saline (10%) Injection for Female Stress Urinary Incontinence and Stress-Predominant Mixed Urinary Incontinence
Brief Title: Hypertonic Saline Injection For Urinary Incontinence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Turgut Ozal University (Other)
Collaborators: Inonu University (Other)
Responsible Party: Principal Investigator, Ibrahim Nuvit Tahtali, Principal Investigator, Turgut Ozal University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6175679-514.04.01-E.28641
Record Dates: First submitted 2021-02-04; First posted 2021-03-23 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Urinary Stress Incontinence
Keywords: Female; Stress Urinary Incontinence; Stress-Predominant Mixed Incontinence; Hypertonic Saline Injection; Therapy
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: This is a single-center prospective before-after (pre-post) interventional study, in which the effectiveness and safety of periurethral hypertonic saline injection were evaluated in female stress urinary incontinence and stress-predominant mixed urinary incontinence patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hypertonic Saline (10%) Injection (Experimental): Periurethral hypertonic saline (10%) injection was performed in female patients with Stress Urinary Incontinence or Stress-Predominant Mixed Urinary Incontinence.
  Interventions: Procedure: Periurethral injection; Drug: Hypertonic (10%) saline

INTERVENTIONS:
Procedure: Periurethral injection — Patients were in the lithotomy position for the procedure. After preparation, topical Lidocaine gel was instilled around the meatus and a 16 F probe was attached. The catheter balloon was inflated to localize the bladder neck and to ensure that injections were performed in the correct anatomical plane. Hypertonic saline (10% NaCl) was injected to the alignment of the urethral meatus in the order of 3-6-9-12 hours of the clock (5 cc to each site, totaling 20 cc). Syringes with 27 Gauge (0.40 mm) outer diameter were used to ensure controlled injection. Since the female urethra is about 4 cm in length, the needle was advanced about 3 cm. Due to the possibility of significant pain with hypertonic saline, 2 cc of Lidocaine hydrochloride was added into the solution.
Drug: Hypertonic (10%) saline — Periurethral hypertonic saline (10%)
  Other Names: 10% NaCl solution

SUMMARY:
The investigators aimed to evaluate the effectiveness and safety of periurethral hypertonic saline (10% NaCl) injection for the treatment of stress urinary incontinence (SUI) and stress-predominant mixed urinary incontinence (MUI) in women.

DETAILED DESCRIPTION:
This single-center prospective pre-post interventional study was conducted between January 2014 and April 2018 with 65 women (44 SUI, 21 MUI). Quality of life was evaluated with the Incontinence Quality of Life Scale (I-QoL) and the lower urinary tract symptoms of women were evaluated with the International Consultation on Incontinence Questionnaire Female Lower Urinary Tract Symptoms Modules (ICIQ-FLUTS). Incontinence status was assessed via the Stamey Incontinence Grade scale. Patients with MUI also were evaluated using the Urinary Distress Inventory-6 (UDI-6). The need for additional treatment (re-injection, other surgical approaches, etc.) was recorded.

Participants were followed up to 24 months after intervention. All outcomes of interest and complications were evaluated/recorded at six preplanned visits (postoperative 1st, 3rd, 6th, 12th, 18th, 24th months).

ELIGIBILITY:
Inclusion Criteria:

The patients who described Stress Urinary Incontinence or Mixed Urinary Incontinence, those who had incontinence during the Valsalva maneuver, patients with positive Marshal-Marchetti test, and those with post-void residual urine volume ≤100 mL were included in the study.

Exclusion Criteria:

Temporary urinary incontinence, delirium, urinary tract infection, urethritis, pure urge incontinence, nocturnal enuresis, decreased bladder compliance and detrusor contraction in the urodynamic study, leakage of urine with low bladder pressure, psychiatric conditions (severe depression and anxiety), body mass index (BMI) >35 kg/m2, and using drugs that may influence bladder storage or emptying

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Change in the Stamey Incontinence Grade at 24 months | Change from baseline at 24 months
  All patients (SUI and MUI) were evaluated as follows: Grade 0: No incontinence; Grade 1: Incontinence with coughing or straining; Grade 2: Incontinence with change in position or walking; Grade 3: Total incontinence at all times
Change in the Urinary Distress Inventory-6 (UDI-6) scores at 1 month | Change from baseline at 1 month
  Only MUI patients were evaluated with UDI-6 scale. UDI-6 is a validated 6-item questionnaire that assesses lower urinary tract symptoms, including incontinence, in women.
Change in the Urinary Distress Inventory-6 (UDI-6) scores at 3 months | Change from baseline at 3 months
  Only MUI patients were evaluated with UDI-6 scale. UDI-6 is a validated 6-item questionnaire that assesses lower urinary tract symptoms, including incontinence, in women.
Change in the Urinary Distress Inventory-6 (UDI-6) scores at 6 months | Change from baseline at 6 months
  Only MUI patients were evaluated with UDI-6 scale. UDI-6 is a validated 6-item questionnaire that assesses lower urinary tract symptoms, including incontinence, in women.
Change in the Urinary Distress Inventory-6 (UDI-6) at 12 months | Change from baseline at 12 months
  Only MUI patients were evaluated with UDI-6 scale. UDI-6 is a validated 6-item questionnaire that assesses lower urinary tract symptoms, including incontinence, in women.
Change in the Urinary Distress Inventory-6 (UDI-6) scores at 18 months | Change from baseline 18 months
  Only MUI patients were evaluated with UDI-6 scale. UDI-6 is a validated 6-item questionnaire that assesses lower urinary tract symptoms, including incontinence, in women.
Change in the Urinary Distress Inventory-6 (UDI-6) scores at 24 months | Change from baseline 24 months
  Only MUI patients were evaluated with UDI-6 scale. UDI-6 is a validated 6-item questionnaire that assesses lower urinary tract symptoms, including incontinence, in women.
Change in the Incontinence Questionnaire Female Lower Urinary Tract Symptoms Modules (ICIQ-FLUTS) scores at 1 month | Change from baseline at 1 month
  All patients (SUI and MUI) were evaluated with the ICIQ-FLUTS which is a questionnaire for evaluating female lower urinary tract symptoms and impact on quality of life of the patients.
Change in the Incontinence Questionnaire Female Lower Urinary Tract Symptoms Modules (ICIQ-FLUTS) scores at 3 months | Change from baseline at 3 months
  All patients (SUI and MUI) were evaluated with the ICIQ-FLUTS which is a questionnaire for evaluating female lower urinary tract symptoms and impact on quality of life of the patients.
Change in the Incontinence Questionnaire Female Lower Urinary Tract Symptoms Modules (ICIQ-FLUTS) scores at 6 months | Change from baseline at 6 months
  All patients (SUI and MUI) were evaluated with the ICIQ-FLUTS which is a questionnaire for evaluating female lower urinary tract symptoms and impact on quality of life of the patients.
Change in the Incontinence Questionnaire Female Lower Urinary Tract Symptoms Modules (ICIQ-FLUTS) scores at 12 months | Change from baseline at 12 months
  All patients (SUI and MUI) were evaluated with the ICIQ-FLUTS which is a questionnaire for evaluating female lower urinary tract symptoms and impact on quality of life of the patients.
Change in the Incontinence Questionnaire Female Lower Urinary Tract Symptoms Modules (ICIQ-FLUTS) scores at 18 months | Change from baseline at 18 months
  All patients (SUI and MUI) were evaluated with the ICIQ-FLUTS which is a questionnaire for evaluating female lower urinary tract symptoms and impact on quality of life of the patients.
Change in the Incontinence Questionnaire Female Lower Urinary Tract Symptoms Modules (ICIQ-FLUTS) scores at 24 months | Change from baseline at 24 months
  All patients (SUI and MUI) were evaluated with the ICIQ-FLUTS which is a questionnaire for evaluating female lower urinary tract symptoms and impact on quality of life of the patients.
Change in the Incontinence Quality of Life Scale (I-QOL) scores at 1 month | Change from baseline at 1 month
  All patients (SUI and MUI) were evaluated with the I-QOL which has 22 questions with the following 3 subscales: avoid and limiting behaviors (items), psychosocial impacts (9 items), and social embarassment (5 items).
Change in the Incontinence Quality of Life Scale (I-QOL) scores at 3 months | Change from baseline at 3 months
  All patients (SUI and MUI) were evaluated with the I-QOL which has 22 questions with the following 3 subscales: avoid and limiting behaviors (items), psychosocial impacts (9 items), and social embarassment (5 items).
Change in the Incontinence Quality of Life Scale (I-QOL) scores at 6 months | Change from baseline at 6 months
  All patients (SUI and MUI) were evaluated with the I-QOL which has 22 questions with the following 3 subscales: avoid and limiting behaviors (items), psychosocial impacts (9 items), and social embarassment (5 items).
Change in the Incontinence Quality of Life Scale (I-QOL) scores at 12 months | Change from baseline at 12 months
  All patients (SUI and MUI) were evaluated with the I-QOL which 22 questions with the following 3 subscales: avoid and limiting behaviors (items), psychosocial impacts (9 items), and social embarassment (5 items).
Change in the Incontinence Quality of Life Scale (I-QOL) scores at 18 months | Change from baseline at 18 months
  All patients (SUI and MUI) were evaluated with the I-QOL which has 22 questions with the following 3 subscales: avoid and limiting behaviors (items), psychosocial impacts (9 items), and social embarassment (5 items).
Change in the Incontinence Quality of Life Scale (I-QOL) scores at 24 months | Change from baseline at 24 months
  All patients (SUI and MUI) were evaluated with the I-QOL which has 22 questions with the following 3 subscales: avoid and limiting behaviors (items), psychosocial impacts (9 items), and social embarassment (5 items).
Need for addtional treatment within the 1st month | Within the 1st month
  Patients who are needed to treat with re-injection or other surgercal approaches.
Need for addtional treatment within 3 months after internvention. | Within the 3 months after internvention.
  Patients who are needed to treat with re-injection or other surgercal approaches.
Need for addtional treatment within 6 months after internvention. | Within the 6 months after internvention.
  Patients who are needed to treat with re-injection or other surgercal approaches.
Need for addtional treatment within 12 months after internvention. | Within the 12 months after internvention.
  Patients who are needed to treat with re-injection or other surgercal approaches.
Need for addtional treatment within 18 months after internvention. | Within the 18 months after internvention.
  Patients who are needed to treat with re-injection or other surgercal approaches.
Need for addtional treatment within 24 months after internvention. | Within the 24 months after internvention.
  Patients who are needed to treat with re-injection or other surgercal approaches.
Presence of complication within 24 months after intervention | Within 24 months after intervention
  Presence of complication such as infection at injection site, urinary tract infection, hematuria, persistent pain, de novo urge incontinence) in all patients.

CONTACTS AND LOCATIONS:
Overall Officials: İbrahim N Tahtali, MD, Principal Investigator — Turgut Ozal University
Locations (2):
- Turkey (Türkiye) (2):
  - Turgut Ozal University, Malatya
  - İnonu University, Malatya

IPD SHARING:
Plan to Share IPD: No
yes

REFERENCES:
- [Background] Irwin GM. Urinary Incontinence. Prim Care. 2019 Jun;46(2):233-242. doi: 10.1016/j.pop.2019.02.004. Epub 2019 Apr 5. PMID 31030824
- [Background] Muth CC. Urinary Incontinence in Women. JAMA. 2017 Oct 24;318(16):1622. doi: 10.1001/jama.2017.15571. No abstract available. PMID 29067430